CLINICAL TRIAL: NCT07294547
Title: Non-Inferiority Assessment of Valacyclovir Versus Valganciclovir as Prophylaxis Against CMV and EBV Viremia in Kidney Transplant Recipients: A Single-Center Prospective Randomized Pilot Study.
Brief Title: Is Valacyclovir Non-inferior to Valganciclovir as CMV and EBV Prophylaxis in Kidney Transplant Recipients? A Single-Center Prospective Randomized Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202507077MINB
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation, Cytomegalovirus Infections; EBV Infection; Antiviral Prophylaxis
Keywords: Non-Inferiority Assessment of Valacyclovir versus Valganciclovir as Prophylaxis Against CMV and EBV Viremia in Kidney Transplant Recipients
MeSH Terms: conditions — Cytomegalovirus Infections; Epstein-Barr Virus Infections | interventions — Valacyclovir; Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Valacyclovir) (Experimental): Standard adult dose for Valacyclovir will be 1000 mg orally twice daily. For pediatric patients, dosing will be weight-based 20 mg/kg/dose twice daily; maximum dose: 1000 mg/dose. The exact dosage will be adjusted for renal function based on published guidelines.
  Patients will continue their assigned prophylactic regimen for at least 6 months.
  Interventions: Drug: Valacyclovir (Valtrex)
- Control group (Valganciclovir) (Active Comparator): Standard adult dose for Valganciclovir will be 450 mg orally once daily. For pediatric patients, dosing will be weight-based 15 mg/kg/dose once daily; maximum dose: 450 mg/dose. The exact dosage will be adjusted for renal function based on published guidelines.
  For pediatric patients who could not swallow pills, Valganciclovir also comes in the form of suspension (prepared by National Taiwan University Hospital in-house pharmacy).
  Patients will continue their assigned prophylactic regimen for at least 6 months.
  Interventions: Drug: Valganciclovir (Valcyte)

INTERVENTIONS:
Drug: Valacyclovir (Valtrex) — Standard adult dose will be 1000 mg orally twice daily. For pediatric patients, dosing will be weight-based 20 mg/kg/dose twice daily; maximum dose: 1000 mg/dose.
  The exact dosage will be adjusted for renal function based on published guidelines.
  Arms: Experimental Group (Valacyclovir)
Drug: Valganciclovir (Valcyte) — Dosing: Standard adult dose will be 450 mg orally once daily. For pediatric patients, dosing will be weight-based 15 mg/kg/dose once daily; maximum dose: 450 mg/dose. The exact dosage will be adjusted for renal function based on published guidelines.
  For pediatric patients who could not swallow pills, Valcyte also comes in the form of suspension (prepared by National Taiwan University Hospital in-house pharmacy).
  Arms: Control group (Valganciclovir)

SUMMARY:
Opportunistic CMV viremia (primary infection or reactivation) is usually managed by taking prophylactic medication for both adult and pediatric kidney transplant patients. Most hospitals prescribe valganciclovir for this purpose but valacyclovir has also been used. The most unfavorable side effect of valganciclovir is bone marrow suppression which can be troublesome for kidney transplant patients who are already immunosuppressed. We aim to assess the non-inferiority of valacyclovir compared with valganciclovir in this study.

DETAILED DESCRIPTION:
CMV viremia and EBV viremia are commonly seen in immunosuppressed kidney transplant recipients. These patients are at highest risk for CMV or EBV viremia early post-transplant or during a period of heightened immunosuppressive regimen to treat acute rejection. CMV viremia could be asymptomatic when the viral load is low, but if uncontrolled, it could lead to severe organ-invasive disease. On the other hand, EBV viremia, though usually not an immediate threat to allograft, harbors risk for post-transplant lymphoproliferative disease (PTLD).Therefore, most transplant centers adopt regular surveillance as well as following certain protocols of antiviral prophylaxis, using valganciclovir specifically against CMV viremia.

Valganciclovir is highly effective as prophylaxis for CMV viremia, but it is also known for its side effects such as myelosuppression and nephrotoxicity. Valacyclovir, though better known for its therapeutic effect for herpes simplex virus, is emerging as an alternative to valganciclovir since some retrospective studies showing its comparative efficacy in CMV prophylaxis. Valacyclovir has favorable side effect profile, and is less expensive. It may also reduce EBV viral shedding in oropharynx, though there's no evidence showing its efficacy in preventing EBV viremia or even PTLD in kidney transplant patients. Given that there are scarce prospective studies comparing these two medications in kidney transplant recipients, our study aims to assess the non-inferiority of valacyclovir compared with valganciclovir as prophylaxis for CMV viremia and investigate its non-inferiority for EBV viremia. We will include both pediatric and adult kidney transplant recipients who received kidney transplant less than 5 years prior to study participation and the patients will be stratified based on their age, years post-transplant, and CMV risk status. Serum viral load and other possible side effects will be monitored during their clinic visits for at least 2 years. The findings from this study will be informative for the design and power calculations for a larger multicenter non-inferiority trial. If valacyclovir is indeed non-inferior to valgancyclovir in both CMV viremia and EBV viremia, utilizing this medication in our post-kidney transplant protocol may help reduce side effect burden and potentially save substantial healthcare cost.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 3 years of age
* Patients who are about to receive or just received kidney transplantation within the past 2 weeks before the date of screening.
* Will be receiving prophylactic antiviral therapy against CMV and/or EBV per discretion of transplant surgeon
* No active CMV or EBV viremia (as defined by detectable viral load PCR) at the time of screening.
* Ability and willingness of the patient (or parent/legal guardian for minors) to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Severe co-morbidities that would preclude safe participation as judged by the transplant surgeon
* Pregnancy (valganciclovir is likely teratogenic)
* Known allergy to both valacyclovir and valganciclovir

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time to new-onset CMV viremia | up to 2 years
Time to new-onset EBV viremia | up to 2 years
Cumulative incidence of new-onset CMV viremia | 6 months, 1year, and 2 years
Cumulative incidence of new-onset EBV viremia | 6 months, 1 year, and 2 years

SECONDARY OUTCOMES:
Bone Marrow Suppression | 6 months, 1 year, 2 years
  The cumulative incidence of specific cytopenia (leukopenia, neutropenia, thrombocytopenia and anemia respectively) in each treatment arm will be compared.
Significantly declined renal function at 2 years post-transplant | 2 years
  The incidence of significant decline in renal function (e.g., >20% decrease from baseline or progression to CKD stage 5) will be compared between groups
Other adverse events during study period | 2 years
  The incidence of other adverse events will be tabulated and compared between groups
Magnitude of Viral Load in New-Onset CMV Viremia | 2 years
  For patients who develop new-onset CMV viremia, the peak CMV viral load (IU/mL) during the viremic episode will be identified.
Magnitude of Viral Load in New-Onset EBV Viremia | 2 years
  For patients who develop new-onset EBV viremia, the peak EBV viral load (IU/mL) during the viremic episode will be identified.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim JS, Lee NR, Park KI, Hwang HS, Lee SH, Chung BH, Jung CW, Cho JH, Park WY, Kim HJ, Jeong JC, Yang J, Lee YH, Park JB, Jeon JS, Lee J, Kim YH, Choi SJN, Oh J, Yoon HE, Kim DG, Shin HS, Ban TH, Kim MS, Ko MJ, Jeong KH; KOTRY study group. Valacyclovir for the prevention of cytomegalovirus infection after kidney transplantation. BMC Infect Dis. 2025 Mar 5;25(1):314. doi: 10.1186/s12879-025-10671-6. PMID 40045190
- [Background] Reischig T, Kacer M, Jindra P, Hes O, Lysak D, Bouda M. Randomized trial of valganciclovir versus valacyclovir prophylaxis for prevention of cytomegalovirus in renal transplantation. Clin J Am Soc Nephrol. 2015 Feb 6;10(2):294-304. doi: 10.2215/CJN.07020714. Epub 2014 Nov 25. PMID 25424991
- [Background] Hoshino Y, Katano H, Zou P, Hohman P, Marques A, Tyring SK, Follmann D, Cohen JI. Long-term administration of valacyclovir reduces the number of Epstein-Barr virus (EBV)-infected B cells but not the number of EBV DNA copies per B cell in healthy volunteers. J Virol. 2009 Nov;83(22):11857-61. doi: 10.1128/JVI.01005-09. Epub 2009 Sep 9. PMID 19740997
- [Background] Cardoso LJC, Martins KAM, Marques PV, Teixeira IPS, Magalhaes E, Minkauskas JL, Faria IC, Ribeiro FM. Valacyclovir versus valganciclovir for cytomegalovirus prophylaxis in kidney transplant recipients: a systematic review and comparative meta-analysis. Clin Transplant Res. 2025 Mar 31;39(1):24-35. doi: 10.4285/ctr.24.0034. Epub 2024 Nov 8. PMID 39510821